CLINICAL TRIAL: NCT06267157
Title: Evaluation of the Effect of the Breastfeeding Counseling Education Model Developed in the Metaverse Universe on the Counseling Skills, Knowledge and Empathy Levels of Nursing Students
Brief Title: Breastfeeding Consultant Training in the Metvaverse Universe
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Sinem Ceylan, Lecturer, Ankara Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023/23
Record Dates: First submitted 2024-01-03; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Feeding
Keywords: Breastfeeding; Metaverse; Nursing; Virtual Reality
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality training (Experimental): Data Collection Forms will be administered face to face to nursing students before training. LactaVerse will be introduced to the students in the experimental group. After the introduction and information are given, virtual reality glasses, lenses and pupil distances will be adjusted and placed on their heads. Each student will be given a disposable goggle mask. Students will then be asked to use their devices in a virtual environment; In the first breastfeeding room, the patient will be asked to touch the entire anatomy, including the breast tissue, ductus, and areola, and examine every angle with the finger. In the next stage; The patient will be asked to go to the second breastfeeding room and assist the mother and baby there. In this room, the student will be expected to complete the skill steps without skipping. He/she will not be able to proceed to the next application without making the correct application.
  Interventions: Device: virtual reality training
- theoretical breastfeeding training (Other): This group will receive 2 hours of theoretical breastfeeding training. Model dolls and breasts will be used in theoretical education by applying the classical education model. Entrance Data Collection Form, Breastfeeding Information Form, Basic Empathy Level Scale, Nursing Counseling Skills Scale and Presence Scale will be applied to the students whose informed consent form has been obtained.
  Interventions: Other: theoretical breastfeeding training

INTERVENTIONS:
Device: virtual reality training — Group that will receive breastfeeding training with virtual glasses, in the metaverse universe.
  Arms: virtual reality training
Other: theoretical breastfeeding training — Classic 2-hour theoretical breastfeeding training with ppt
  Arms: theoretical breastfeeding training

SUMMARY:
Although breastfeeding is an important and natural process in infant development, mothers may fail to manage the process. Nurses, who have an important place in helping to physically initiate and maintain breastfeeding, provide an in-depth knowledge of breast anatomy and breastfeeding physiology, practice and process breastfeeding techniques. Must have extensive management skills. Although the World Health Organization recommends that breastfeeding issues should be addressed in medical, nursing and midwifery schools, there is a lack of nurses' training curricula and breastfeeding training given in hospitals. Due to this deficiency, mothers have low self-confidence and insufficient knowledge about breastfeeding.

The aim of this project is to develop a breastfeeding counseling model in the metaverse universe and to determine the effect of this model on nursing students' breastfeeding counseling skills, knowledge level and empathy skills. Giving breastfeeding education with the metaverse application compared to the application on real patients includes much less risk for the patient and the ability to practice until the right skill is acquired. In the project, it is expected that the breastfeeding counseling education model (LactaVerse), which is structured on virtual reality developed in the metaverse universe, is compared to the existing deficient and non-standardized breastfeeding education practice, enabling nurses to practice more and without errors during the undergraduate education, and to gain more effective skills in breastfeeding counseling. In this context, the project will support the ability of multiple users in the metaverse universe to examine the anatomy of the breast and apply breastfeeding counseling to the mother by transmitting their voices and movements with virtual glasses.

In the preparation phase of the training to be developed in the virtual universe within the scope of the project, the breast anatomical modeling and the breastfeeding mother-baby duo project scenario will be developed and virtual glasses will be transferred. At this stage, expert opinions of the questionnaires to be used in the evaluation of educational effectiveness will be taken. Pre-application of data collection tools and LactaVerse training will be made. Experiment (n=40) and control (n=40) groups will be determined from the students by randomization. "Descriptive Characteristics Data Collection Form", "Breastfeeding Information Form", "Basic Empathy Level Scale", "Nursing Counseling Skill Scale" and "Presence Scale" will be applied to both groups. During the application phase, Lactaverse training method with virtual glasses will be applied to the experimental group, and a 2-hour theoretical classical training method will be applied to the control group. After 4 weeks of the training, the post-tests will be applied to the experimental group and the control group and they counseling will be given to the patient who plays the role of a nursing mother in the laboratory, and measurements will be made with the Breastfeeding Counseling Skill List and statistical analyzes will be applied.

With the training developed in connection with the project, it is expected that nurses will have a high level of empathy development and breastfeeding counseling skills in a complex healthcare environment such as breastfeeding counseling before they graduate. In this way, the professional knowledge, counseling skills and empathy skills of nurses, who have an important role in breastfeeding, will increase, helping our society to increase the breastfeeding rates to the desired level.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Not having received formal training on breastfeeding
* No vision or hearing problems
* Not having a motion sensitive disease (e.g. Vertigo).

Exclusion Criteria:

* Withdrawing from the research voluntarily
* Not participating in the stages of the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-07-02 (Estimated)

PRIMARY OUTCOMES:
Introductory Features Data Collection Form | 5 mounth
  The form prepared by the researchers consists of 2 parts and a total of 13 questions. In the first part, there are 8 questions about the socio-demographic characteristics of the students, and in the second part, there are 5 questions questioning their computer game playing situations and virtual reality application experiences.
Breastfeeding Information Form | 5 mounth
  This form consists of 25 questions to be answered as true, false and unknown in 5 subgroups. Each correct answer is worth 4 points, with the highest 100 and the lowest 0 points. As the score obtained from the form increases, the level of breastfeeding knowledge will be interpreted as increasing. After the preparation of this form, it was revised by taking expert opinions from 10 faculty members working in the field. The reliability of the information form will be measured by the Kuder Richardson 20 (KR-20) test.
Basic Empathy Level Scale | 5 mounth
  This scale is a 5-point Likert-type graded, two-factor, and 20-item scale. It consists of a total of 20 items, 9 items measure cognitive empathy and 11 items measure emotional empathyFor the cognitive empathy subscale, the lowest score that can be obtained from the scale is 9 and the highest score is 45. For the emotional empathy subscale, the lowest score that can be obtained from the scale is 11 and the highest score is 55. Since there is no cut-off point in the scale scoring, it is used in comparison studies. The higher the score obtained from the scale determines the higher the basic empathy level.
Breastfeeding Teaching Skill Evaluation Form | 5 mounth
  It will be scored on whether the student doing the breastfeeding counseling is able to demonstrate the skill. There are 25 digits in the Skill List.
  Correct application will be evaluated as 2, incomplete application will be evaluated as 1, inability to apply will be evaluated as 0 points, and the maximum score to be obtained from the list is 50 and the minimum score is 0.
Presence Scale | 5 mounth
  his scale has 5 sub-dimensions and 5-point Likert type. The sub-dimensions of the scale were determined as Participation, Adaptation/Containment, Sensory Commitment, Interaction and Interface Quality. It is assumed that as the scores obtained from the sub-dimensions increase, the experienced virtual environment is perceived in a more realistic structure and the sense of presence is at a higher level.

CONTACTS AND LOCATIONS:
Overall Officials: Gülten Güvenc, Study Director
Locations (1):
- Gulhane Faculty of Nursing, Ankara, Turkey (Türkiye)